CLINICAL TRIAL: NCT03632733
Title: Effects of Antimicrobials on the Altered Skin Flora in Patients With Palmar Arsenical Keratosis
Brief Title: Effects of Antimicrobials on the Altered Skin Flora in Arsenical Keratosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Asiya Ferdous, Resident, Department of Pharmacology, BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.BSMMU/2018/924
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Keratotic Nodular Size
MeSH Terms: interventions — Tetracycline; Clotrimazole

STUDY DESIGN:
Intervention Model Description: Three antimicrobials ( two single and one in combination form) and a placebo will be provided in patients randomly
Who Masked: Participant
Masking Description: Participants are not aware of the drug they are given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tetracycline group (Active Comparator): Tetracycline cream twice daily for three months
  Interventions: Drug: Tetracycline
- Clotrimazole group (Active Comparator): Clotrimazole cream twice daily for three months
  Interventions: Drug: Clotrimazole
- Combination drug group (Active Comparator): Tetracycline and Clotrimazole combination cream twice daily for three months
  Interventions: Drug: Tetracycline and Clotrimazole
- Placebo group (Placebo Comparator): participants will be provided a cream containing no active drug ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tetracycline — Tetracycline cream
  Other Names: Tetrax
  Arms: Tetracycline group
Drug: Clotrimazole — Clotrimazole cream
  Other Names: Clotrim
  Arms: Clotrimazole group
Drug: Tetracycline and Clotrimazole — Combination cream
  Other Names: No other name
  Arms: Combination drug group
Other: Placebo — Placebo cream without active drug ingredients
  Other Names: No other name
  Arms: Placebo group

SUMMARY:
It had been found in certain studies that there is an alteration of normal skin flora in patients with arsenical keratosis. The relationship between such altered skin flora and development of keratosis in arsenicosis is not established or explored.There is no such study where effects of antimicrobials have been evaluated as the treatment of arsenical keratosis. So the present study is designed to see the effects of antimicrobials on the altered skin flora (Enterobacter and Aspergillus) in patients with palmar arsenical keratosis.

DETAILED DESCRIPTION:
According to a working group of World Health Organization, arsenicosis is a chronic health condition arising from prolonged ingestion (not less than six months) of arsenic above a safe level, usually manifested by characteristic and most diagnostic skin lesions, like- melanosis, leucomelanosis and keratosis, with or without involvement of internal organs. Arsenical keratosis usually appears on palm of the hand and plantar aspect of the feet and may also develop on the dorsum of the extremities and trunk. It had been found in certain studies that there is an alteration of normal skin flora in patients with arsenical keratosis. The relationship between such altered skin flora and development of keratosis in arsenicosis is not established or explored. Treatment of all types of keratosis is difficult. The most common therapeutic option leads to short-term improvement and is frequently associated with various adverse effects. Treatment tends to be symptomatic and includes topical keratolytic, orally administered antioxidant vitamins and minerals, or reconstructive surgery with total excision of the keratotic skin followed by grafting. There is no such study where effects of antimicrobials have been evaluated as the treatment of arsenical keratosis. So the present study is designed to see the effects of antimicrobials on the altered skin flora (Enterobacter and Aspergillus) in patients with palmar arsenical keratosis. The present study will be a clinical trial. The study will take place at the Department of Pharmacology, Department of Microbiology and Immunology of Bangabandhu Sheikh Mujib Medical University and at Laksham Upazilla of Comilla District from September 2017 to February 2019. After including participants as per selection criteria, written informed consent will be taken from all of them. Then water, nail, skin swab and scrapping samples will be collected and analyzed in the laboratory. After doing culture sensitivity, antimicrobials will be given to the patients. The duration of treatment will be decided upon sensitive drugs. Keratotic nodular size will be measured of each patient to draw a conclusion about the effect of antimicrobials in patients with palmar arsenical keratosis. As it had been found in previous studies conducted at the Department of Pharmacology of Bangabandhu Sheikh Mujib Medical University that both skin bacterial and fungal flora were altered in patients with arsenical keratosis, this study will be done to establish the relationship between such alteration and arsenical keratosis by exploring the effects of antimicrobials as a treatment of keratosis.

ELIGIBILITY:
Inclusion Criteria:

Drinking arsenic contaminated water (>50 microgram/ litre) for more than 6 months

Patient with moderate to severe arsenical palmar keratosis

Patient voluntarily agreed to participate

Patient did not receive topical application of any drug for the last three months

Patient who understood the instructions of applying drug and could apply drug as per as instructions -

Exclusion Criteria:

Patient who received any treatment of arsenicosis within last three months

Patient with diagnosed skin diseases, like- atopic dermatitis and psoriasis

Any diagnosed systemic diseases, inflammatory disease and infectious condition that affect the skin, for example- diabetes melitus, SLE and hepatitis

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in keratotic nodular size | three months
  palmar arsenical keratosis will be measured before and after applying interventions

CONTACTS AND LOCATIONS:
Overall Officials: Asiya Ferdous, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Eruain Community Clinic, Lākshām, Bangladesh